CLINICAL TRIAL: NCT00754455
Title: A Phase 2a Randomized, Double Blind, Placebo Controlled Trial to Evaluate the Safety and Immunogenicity of a Seasonal Influenza Virus-Like Particle (VLP) Vaccine (Recombinant) in Healthy Adults
Brief Title: Evaluate the Safety and Immunogenicity of a Seasonal Influenza VLP Vaccine (Recombinant) in Healthy Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novavax (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: NVX 755.201
Record Dates: First submitted 2008-09-16; First posted 2008-09-18 (Estimated); Last update posted 2013-07-18 (Estimated); Status verified 2013-07

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Low dose (Experimental)
  Interventions: Biological: Influenza VLP Vaccine (recombinant)
- Mid dose (Experimental)
  Interventions: Biological: Influenza VLP Vaccine (recombinant)
- High dose (Experimental)
  Interventions: Biological: Influenza VLP Vaccine (recombinant)
- Placebo (Placebo Comparator)
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Influenza VLP Vaccine (recombinant) — Single injection Day 0; 0.5mL
  Arms: High dose; Low dose; Mid dose
Biological: Placebo — Placebo as a single injection of 0.5 mL.
  Arms: Placebo

SUMMARY:
A Phase 2a Randomized, Double Blind, Placebo Controlled Trial to Evaluate the Safety and Immunogenicity of a Seasonal Influenza Virus-Like Particle (VLP) Vaccine (recombinant) in Healthy Adults.

Study Objectives:

Primary:

* To assess the tolerability and safety of Influenza VLP Vaccine
* To assess the immunogenicity of Influenza VLP Vaccine as measured by hemagglutination inhibition (HAI) antibody titers to each of the three component viral strains

Secondary:

* To evaluate the cross-strain immunogenicity of Influenza VLP Vaccine as measured by hemagglutination inhibition (HAI) antibody titers against drifted strains
* To quantify antibody against neuraminidase and hemagglutinin following administration of Influenza VLP Vaccine
* To assess cell-mediated immune (CMI) responses to Influenza VLP Vaccine as quantified by interferon-gamma (IFNg) and Granzyme-B produced by peripheral blood mononuclear cells (PBMCs).

DETAILED DESCRIPTION:
Study Design:

This is a Phase 2a randomized, double-blind, placebo-controlled study to evaluate the safety, tolerability and immunogenicity of three dose levels (low, middle or high) of Influenza VLP Vaccine or placebo in healthy adults(18 to 49 years of age).

Eligible subjects will provide a blood sample for baseline evaluation of immunological measures followed by a single intramuscular (IM) injection of Influenza VLP Vaccine or placebo (Day 1).

Subjects will be monitored in the clinic for a period of at least 30 minutes following vaccination for the occurrence of adverse events including local injection site reactions and systemic responses. For 7 days following vaccination and beginning the day of vaccination, subjects will maintain a symptom diary for daily recording of injection-site reactions as well as generalized systemic reactions including measurement of body temperature. Clinic staff will contact the subjects by telephone 2 days post vaccination (Day 3) to check for adverse events and to answer any questions related to collection of symptom diary information. Subjects will return to the clinic 7 days following vaccination (Day 8) for safety evaluation that will include a review of diary card information. A subset of subjects will additionally return to the clinic 10-14 days following vaccination (Days 11-15) to provide a blood sample for evaluation of cell-mediated immune (CMI) responses. All subjects will return to the clinic 21 days following injection (Day 22) for a safety evaluation and to provide a blood sample for measurement of humoral immunological parameters. A final safety evaluation (telephone contact) will occur at approximately 6 months following vaccination (Day 181).

The study will be conducted as a parallel group design with a total of approximately 300 subjects (18 to 49 years of age) randomly assigned to one of 4 treatment arms (high, middle, low and placebo) in a 2:2:1:1 ratio. The following is a summary of subject allocation to treatment:

Subject Allocation Treatment Condition Number of Subjects High dose vaccine/ 0.5 mL - 100 Middle dose vaccine/ 0.5 mL - 100 Low dose vaccine/ 0.5 mL - 50 Placebo (0.5 mL) - 50

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female 18 to 49 years of age at the time of the vaccination.
2. Informed consent must be obtained from the subject prior to beginning any study specific procedures indicating that they understand the purpose of this study and are willing to adhere to the procedures described in this protocol.
3. Available by telephone.
4. Free of obvious health problems or chronic illnesses (i.e., recent exacerbation or acute episode of chronic illness in the last 3 months) as established by medical history, review of systems and clinical examination before entering the study. This includes any mental condition that would interfere with subject self-assessment. Subjects with pre-existing stable disease, defined as no significant disease diagnosed in the month prior to study vaccine receipt and disease not requiring significant change in therapy or hospitalization for worsening disease 3 months before receipt of study vaccine are eligible.
5. If subject is of childbearing potential, she must be abstinent or have used adequate contraceptive precautions (e.g., intrauterine contraceptive device; oral contraceptives or other equivalent hormonal contraception) for 3 months prior to vaccination. She must also have a negative pregnancy test at study entry and must agree to continue such precautions for three months after vaccination.

Exclusion Criteria:

1. Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine(s) within 30 days preceding the administration of the study vaccine, or planned use during the study period.
2. Has received any other licensed vaccines within 4 weeks prior to enrollment in this study or expected receipt of any vaccination before the final immune response blood collection.
3. Has received any influenza vaccine within the prior 6 month period.
4. Chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying drugs within six months prior to the administration of the study vaccine. The use of inhaled and nasal steroids will be permitted.
5. Any medically diagnosed or suspected immunodeficient condition based on medical history and physical examination.
6. Administration of immunoglobulins and/or any blood products within the three months preceding the administration of the study vaccine or during the study.
7. Acute disease at the time of enrollment. Acute disease is defined as the presence of a moderate or severe illness with or without fever ≥ 100.5º F.
8. Acute clinically significant pulmonary, cardiovascular, hepatic or renal functional abnormality, as determined by physical examination or laboratory screening tests.
9. Major congenital defects or serious chronic illness.
10. History of any neurological disorders or seizures, with the exception of febrile seizures during childhood.
11. Pregnant or lactating female.
12. Females planning to become pregnant or planning to discontinue contraceptive precautions within 60 days of enrollment in this study.
13. Any condition that in the opinion of the investigator would interfere with evaluation of the vaccine or interpretation of study results.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 317 (Actual)
Dates: Start 2008-09; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
To assess the tolerability and safety of Influenza VLP Vaccine | 6 Months
To assess the immunogenicity of Influenza VLP Vaccine as measured by hemagglutination inhibition (HAI) antibody titers to each of the component viral strains | Day 22

SECONDARY OUTCOMES:
To evaluate cross-strain immunogenicity as measured by HAI titers against drifted strains | Day 22
To quantify antibody responses against neuraminidase and hemagglutinin | Day 22
To assess cell-mediated immune (CMI) responses to Influenza VLP Vaccine | Day 11

CONTACTS AND LOCATIONS:
Overall Officials: John E Ervin, M.D., Principal Investigator — The Center for Pharmaceutical Research; Laurence Chu, M.D., Principal Investigator — Benchmark Research; Larry Gilderman, D.O., Principal Investigator — University Clinical Research; David L Freid, M.D., Principal Investigator — Omega Medical Research
Locations (4):
- United States (4):
  - University Clinical Research, Pembroke Pines, Florida
  - The Center for Pharmacuetical Research, Kansas City, Missouri
  - Omega Medical Research, Warwick, Rhode Island
  - Benchmark Research, Austin, Texas